CLINICAL TRIAL: NCT01410747
Title: Specified Drug Use-Results Survey on Long-Term Treatment for Prograf® Capsules 0.5 mg, 1 mg Lupus Nephritis
Brief Title: A Study to Evaluate the Safety and Efficacy of Tacrolimus for Lupus Nephritis Under Actual Use Situations
Acronym: TRUST
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PRGN01
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2020-03

CONDITIONS: Lupus Nephritis
Keywords: long-term treatment; tacrolimus; renal failure
MeSH Terms: conditions — Lupus Nephritis; Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tacrolimus group: Oral
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: FK506

SUMMARY:
To evaluate the safety and efficacy of tacrolimus for lupus nephritis under actual-use.

DETAILED DESCRIPTION:
The objectives of the survey are to evaluate the safety and efficacy of tacrolimus for lupus nephritis under actual-use situations, and to identify factors that might affect the safety and efficacy of tacrolimus. In addition, long-term renal outcome will be evaluated.

ELIGIBILITY:
patients receiving tacrolimus for the treatment of lupus nephritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients receiving tacrolimus for the treatment of lupus nephritis
Sampling Method: Non-Probability Sample
Enrollment: 1484 (Actual)
Dates: Start 2007-04-10 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of renal events (renal failure and progression to dialysis) | Up to 10 years

SECONDARY OUTCOMES:
24-hour urinary protein | Baseline, 4 week, 8 week, 12 week, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year, 9 year, 10 year
Urinary red blood cell (RBC) count | Baseline, 4 week, 8 week, 12 week, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year, 9 year, 10 year
Serum creatinine | Baseline, 4 week, 8 week, 12 week, 1 year, 2 year, 3 year, 4 year, 5 year, 6 year, 7 year, 8 year, 9 year, 10 year

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Shagoku
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Takeuchi T, Wakasugi N, Hashida T, Uno S, Makino H. Long-Term Safety and Effectiveness of Tacrolimus in Patients With Lupus Nephritis in Japan: 10-Year Analysis of the Real-World TRUST Study. J Rheumatol. 2024 Jun 1;51(6):613-621. doi: 10.3899/jrheum.2023-0210. PMID 38359944
- [Derived] Takeuchi T, Wakasugi N, Uno S, Makino H. Long-term Safety and Effectiveness of Tacrolimus in Patients With Lupus Nephritis: 5-year Interim Postmarketing Surveillance Study in Japan (TRUST). J Rheumatol. 2021 Jan 1;48(1):74-81. doi: 10.3899/jrheum.191008. Epub 2020 Apr 1. PMID 32238515